CLINICAL TRIAL: NCT05900154
Title: A PHASE 1, OPEN-LABEL, AGE-DESCENDING, DOSE-FINDING STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF RESPIRATORY SYNCYTIAL VIRUS PREFUSION F SUBUNIT VACCINE (RSVpreF) IN CHILDREN 2 TO <18 YEARS OF AGE
Brief Title: A Study to Learn About the Safety and Immune Activity of RSVpreF in Children 2 to <18 Years of Age
Acronym: PICASSO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: C3671016; 2024-000422-17 (EudraCT Number)
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: RESPIRATORY SYNCYTIAL VIRUS (RSV)
Keywords: RESPIRATORY SYNCYTIAL VIRUS; RSV; RSV vaccine; Respiratory illness; Respiratory infection; Pediatric
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: This is an open-label dose-finding study. A single dose of RSVpreF 120 µg will be given to 40 participants in the 5 to <18 age group first. Upon safety review and approval, a dose of 60 µg will be given to 20 participants in the 2 to <5 age group. If, 60 µg is safe, another 20 participants in the 2 to <5- age group will receive the 120-µg dose. Approximately 60 to 120 participants are expected to be enrolled.
Masking Description: This study is open-label therefore no blinding requirements are in place since all participants will receive RSVPreF.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- standard dose in 5 to <18 years olds, healthy (Experimental): standard dose (120 µg)
  Interventions: Biological: RSVpreF 120 µg
- standard dose in 5 to < 18 years olds, with chronic high risk conditions (Experimental): standard dose (120 µg)
  Interventions: Biological: RSVpreF 120 µg
- standard dose in 2 to < 5 years olds (Experimental): standard dose (120 µg)
  Interventions: Biological: RSVpreF 120 µg
- low dose in 5 to <18 years olds, healthy (Experimental): low dose (60 µg)
  Interventions: Biological: RSVpreF 60 µg
- low dose in 5 to <18 years olds, with chronic high risk conditions (Experimental): low dose (60 µg)
  Interventions: Biological: RSVpreF 60 µg
- low dose in 2 to < 5 years olds (Experimental): low dose (60 µg)
  Interventions: Biological: RSVpreF 60 µg

INTERVENTIONS:
Biological: RSVpreF 120 µg — RSVpreF standard dose level
  Arms: standard dose in 2 to < 5 years olds; standard dose in 5 to < 18 years olds, with chronic high risk conditions; standard dose in 5 to <18 years olds, healthy
Biological: RSVpreF 60 µg — RSVpreF low dose level
  Arms: low dose in 2 to < 5 years olds; low dose in 5 to <18 years olds, healthy; low dose in 5 to <18 years olds, with chronic high risk conditions

SUMMARY:
The purpose of this study is to learn about the safety and immune activity of the vaccine (called RSVpreF) in children 2 to <18 years of age.

This study will identify the dose level to be used in Phase 2/3 trials in this age cohort. All participants will receive one injection of RSVpreF. This study has four study visits, two in-clinic and two telehealth visits. Blood samples will be collected for testing. This study is about 6 months long for each participant and will be conducted in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Participants 2 to <18 years of age at enrollment
2. Participants 2 to <18 years of age should either be healthy or be considered by the investigator to be at high risk of RSV disease based on the presence of 1 of the following chronic medical conditions:

   * Cystic fibrosis
   * Medically treated asthma
   * Other chronic respiratory diseases and malformations of the lung
   * Down syndrome
   * Neuromuscular disease
   * Cerebral palsy
   * Hemodynamically significant or symptomatic congenital heart disease
3. All participants 2 to <5 years of age must be seropositive for RSV as confirmed by serology.
4. Participants' parent(s)/legal guardian(s) and participants, as age appropriate, who are willing and able to comply with all scheduled visits, investigational plan, laboratory tests, and other study procedures, including collection of nasal swabs by participants' parent(s)/legal guardian(s) and by study staff when indicated.
5. The participant's parent(s)/legal guardian is capable of giving signed informed consent as described in the protocol. Depending on the age of the participant and according to local requirements, participants will also be asked to provide assent as appropriate (verbal or written).

Exclusion Criteria:

1. Immunocompromised individuals associated with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
2. Individuals with a history of autoimmune disease or an active autoimmune disease requiring therapeutic intervention, including but not limited to systemic lupus erythematosus. Note: Stable type 1 diabetes and hypothyroidism are permitted.
3. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
4. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
5. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
6. Individuals with a history of epilepsy or other seizure disorders, or a history of seizures and/or other neurological complications following vaccination.
7. Previous vaccination with any licensed or investigational RSV vaccine or planned receipt during study participation. Children who may have been exposed to investigational RSV vaccines through maternal immunization will be permitted.
8. Receipt of investigational or approved monoclonal antibodies against RSV within 6 months before study intervention administration, or planned receipt throughout the study.
9. Receipt of blood/plasma products or immunoglobulins within 28 days before study intervention administration, or planned receipt throughout the study.
10. Receipt of chronic systemic treatment with known immunosuppressant medications (including cytotoxic agents or systemic corticosteroids), or radiotherapy, within 60 days before study intervention administration, or planned receipt throughout the study.

    Note: Systemic corticosteroids are defined as those administered for ≥14 days at a dose of ≥20 mg/day of prednisone or equivalent (eg, for cancer or an autoimmune disease). Inhaled/nebulized, intra-articular, intrabursal, or topical (skin, eyes, or ears) corticosteroids are permitted.
11. Participation in other studies involving study intervention within 28 days prior to study entry and/or for the duration of study participation.
12. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- United States (17):
  - University of Alabama at Birmingham - School of Medicine, Birmingham, Alabama
  - Stanford University Medical Center, Palo Alto, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Bio-Medical Research LLC, Miami, Florida
  - Velocity Clinical Research, Sioux City, Sioux City, Iowa
  - Velocity Clinical Research, New Orleans, Metairie, Louisiana
  - Velocity Clinical Research, Omaha, Omaha, Nebraska
  - Rochester Clinical Research, LLC, Rochester, New York
  - Duke Vaccine And Trials Unit, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Senders Pediatrics, South Euclid, Ohio
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Innovo Research - Austin Regional Clinic, Austin, Texas
  - Velocity Clinical Research, Austin, Austin, Texas
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Seattle Children's - Building Cure, Seattle, Washington
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3671016

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 128 participants were enrolled, however 1 participant was assigned to a vaccine group but did not receive vaccination. Consequently, a total of 127 participants were vaccinated.
Pre-assignment Details: Participants were divided into 2 age groups: 5 to less than (<) 18 years and 2 to < 5 years. Participants in 5 to <18 years age group were further stratified as healthy and with high-risk chronic medical conditions.
Groups:
- RSVpreF 120 Micrograms (mcg): 5 to <18 Years [Healthy Participants]: Healthy participants of age 5 to <18 years received a single dose of respiratory syncytial virus stabilized prefusion F subunit vaccine (RSVpreF) 120 mcg intramuscularly on Day 1.
- RSVpreF 120 mcg: 5 to <18 Years [High Risk Participants]: Participants who had high risk chronic medical conditions of age 5 to <18 years received a single dose of RSVpreF 120 mcg intramuscularly on Day 1.
- RSVpreF 120 mcg: 2 to < 5 Years: Participants of age 2 to <5 years received a single dose of RSVpreF 120 mcg intramuscularly on Day 1.
- RSVpreF 60 mcg: 5 to <18 Years [Healthy Participants]: Healthy participants of age 5 to <18 years received a single dose of RSVpreF 60 mcg intramuscularly on Day 1.
- RSVpreF 60 mcg: 5 to <18 Years [High Risk Participants]: Participants who had high risk chronic medical conditions of age 5 to <18 years received a single dose of RSVpreF 60 mcg intramuscularly on Day 1.
- RSVpreF 60 mcg: 2 to < 5 Years: Participants of age 2 to <5 years received a single dose of RSVpreF 60 mcg intramuscularly on Day 1.
Period: Vaccination Period
Arm/Group | RSVpreF 120 Micrograms (mcg): 5 to <18 Years [Healthy Participants] | RSVpreF 120 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 120 mcg: 2 to < 5 Years | RSVpreF 60 mcg: 5 to <18 Years [Healthy Participants] | RSVpreF 60 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 60 mcg: 2 to < 5 Years
Started | 25 | 23 | 24 | 17 | 18 | 20
Completed | 25 | 23 | 24 | 17 | 18 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Follow-Up Period
Arm/Group | RSVpreF 120 Micrograms (mcg): 5 to <18 Years [Healthy Participants] | RSVpreF 120 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 120 mcg: 2 to < 5 Years | RSVpreF 60 mcg: 5 to <18 Years [Healthy Participants] | RSVpreF 60 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 60 mcg: 2 to < 5 Years
Started | 25 | 23 | 24 | 17 | 18 | 20
Completed | 24 | 21 | 23 | 17 | 17 | 19
Not Completed | 1 | 2 | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 2 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who received the study intervention.
Groups:
- RSVpreF 120 mcg: 5 to <18 Years [Healthy Participants]: Healthy participants of age 5 to <18 years received a single dose of RSVpreF 120 mcg intramuscularly on Day 1.
- Total: Total of all reporting groups
Arm/Group | RSVpreF 120 mcg: 5 to <18 Years [Healthy Participants] | RSVpreF 120 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 120 mcg: 2 to < 5 Years | RSVpreF 60 mcg: 5 to <18 Years [Healthy Participants] | RSVpreF 60 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 60 mcg: 2 to < 5 Years | Total
Number analyzed (Participants) | 25 | 23 | 24 | 17 | 18 | 20 | 127
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 9 | 11 | 24 | 12 | 12 | 20 | 88
  Adolescents (12-17 years) | 16 | 12 | 0 | 5 | 6 | 0 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 13 | 5 | 7 | 7 | 58
  Male | 10 | 12 | 11 | 12 | 11 | 13 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 1 | 3 | 4 | 5 | 18
  Not Hispanic or Latino | 20 | 23 | 22 | 14 | 13 | 15 | 107
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 6 | 3 | 2 | 6 | 4 | 28
  White | 16 | 17 | 17 | 13 | 9 | 15 | 87
  More than one race | 0 | 0 | 3 | 2 | 3 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Vaccination
Description: Local reactions were collected in the electronic diary (e-diary) from Day 1 through Day 7 after vaccination. Local reactions included pain at injection site, redness, and swelling. For participants greater than or equal to (>=) 2 years to <12 years of age, redness and swelling were graded as mild: 0.5 to 2.0 centimeter (cm), moderate: >2.0 to 7.0 cm, and severe: > 7 cm; for participants >=12 years of age, mild: > 2.0 to 5.0 cm, moderate: >5.0 to 10.0 cm, and severe: >10 cm. Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), and severe (prevented daily activity).
Time Frame: Day 1 through Day 7 after Vaccination
Population: Safety population included all enrolled participants who received study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- RSVpreF 120 mcg: 2 to <5 Years: Participants of age 2 to <5 years received a single dose of RSVpreF 120 mcg intramuscularly on Day 1.
- RSVpreF 60 mcg: 2 to <5 Years: Participants of age 2 to <5 years received a single dose of RSVpreF 60 mcg intramuscularly on Day 1.
Arm/Group | RSVpreF 120 mcg: 5 to <18 Years [Healthy Participants] | RSVpreF 120 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 120 mcg: 2 to <5 Years | RSVpreF 60 mcg: 5 to <18 Years [Healthy Participants] | RSVpreF 60 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 60 mcg: 2 to <5 Years
Number analyzed (Participants) | 25 | 23 | 24 | 17 | 18 | 20
Percentage of participants
  Pain at injection site: Mild | 36.0 [18.0 to 57.5] | 39.1 [19.7 to 61.5] | 8.3 [1.0 to 27.0] | 35.3 [14.2 to 61.7] | 33.3 [13.3 to 59.0] | 15.0 [3.2 to 37.9]
  Pain at injection site: Moderate | 8.0 [1.0 to 26.0] | 8.7 [1.1 to 28.0] | 0 [0.0 to 14.2] | 5.9 [0.1 to 28.7] | 22.2 [6.4 to 47.6] | 0 [0.0 to 16.8]
  Pain at injection site: Severe | 4.0 [0.1 to 20.4] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 19.5] | 0 [0.0 to 18.5] | 0 [0.0 to 16.8]
  Redness: Mild | 12.0 [2.5 to 31.2] | 4.3 [0.1 to 21.9] | 12.5 [2.7 to 32.4] | 0 [0.0 to 19.5] | 11.1 [1.4 to 34.7] | 5.0 [0.1 to 24.9]
  Redness: Moderate | 12.0 [2.5 to 31.2] | 4.3 [0.1 to 21.9] | 0 [0.0 to 14.2] | 5.9 [0.1 to 28.7] | 0 [0.0 to 18.5] | 0 [0.0 to 16.8]
  Redness: Severe | 0 [0.0 to 13.7] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 19.5] | 0 [0.0 to 18.5] | 0 [0.0 to 16.8]
  Swelling: Mild | 4.0 [0.1 to 20.4] | 0 [0.0 to 14.8] | 4.2 [0.1 to 21.1] | 0 [0.0 to 19.5] | 11.1 [1.4 to 34.7] | 0 [0.0 to 16.8]
  Swelling: Moderate | 8.0 [1.0 to 26.0] | 8.7 [1.1 to 28.0] | 0 [0.0 to 14.2] | 5.9 [0.1 to 28.7] | 11.1 [1.4 to 34.7] | 5.0 [0.1 to 24.9]
  Swelling: Severe | 0 [0.0 to 13.7] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 19.5] | 0 [0.0 to 18.5] | 0 [0.0 to 16.8]

2. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination
Description: Systemic events included fever, fatigue, headache, vomiting, diarrhea, muscle pain and joint pain and were recorded by participants using e-diary. Fever: oral temperature >= 38.0 degree Celsius (deg C) and categorized as >=38.0 to 38.4 deg C (mild), >38.4 to 38.9 deg C (moderate), and >38.9 to 40.0 deg C (severe). Fatigue, headache, muscle pain and joint pain were graded as mild (did not interfere with activity), moderate (some interference with activity), and severe (prevented daily routine activity). Vomiting was graded mild: 1-2 times in 24 hours (h), moderate: >2 times in 24h, and severe: required intravenous hydration. Diarrhea was graded mild: 2-3 loose stools in 24h, moderate: 4-5 loose stools in 24h and severe: 6 or more loose stools in 24h.
Time Frame: Day 1 through Day 7 after Vaccination
Population: Safety population included all enrolled participants who received study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSVpreF 120 mcg: 5 to <18 Years [Healthy Participants] | RSVpreF 120 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 120 mcg: 2 to <5 Years | RSVpreF 60 mcg: 5 to <18 Years [Healthy Participants] | RSVpreF 60 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 60 mcg: 2 to < 5 Years
Number analyzed (Participants) | 25 | 23 | 24 | 17 | 18 | 20
Percentage of participants
  Fever: Mild | 0 [0.0 to 13.7] | 4.3 [0.1 to 21.9] | 4.2 [0.1 to 21.1] | 0 [0.0 to 19.5] | 0 [0.0 to 18.5] | 5.0 [0.1 to 24.9]
  Fever: Moderate | 0 [0.0 to 13.7] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 19.5] | 5.6 [0.1 to 27.3] | 0 [0.0 to 16.8]
  Fever: Severe | 0 [0.0 to 13.7] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 5.9 [0.1 to 28.7] | 5.6 [0.1 to 27.3] | 0 [0.0 to 16.8]
  Fatigue: Mild | 20.0 [6.8 to 40.7] | 21.7 [7.5 to 43.7] | 20.8 [7.1 to 42.2] | 41.2 [18.4 to 67.1] | 16.7 [3.6 to 41.4] | 30.0 [11.9 to 54.3]
  Fatigue: Moderate | 12.0 [2.5 to 31.2] | 21.7 [7.5 to 43.7] | 8.3 [1.0 to 27.0] | 5.9 [0.1 to 28.7] | 33.3 [13.3 to 59.0] | 5.0 [0.1 to 24.9]
  Fatigue: Severe | 0 [0.0 to 13.7] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 19.5] | 0 [0.0 to 18.5] | 0 [0.0 to 16.8]
  Headache: Mild | 16.0 [4.5 to 36.1] | 26.1 [10.2 to 48.4] | 0 [0.0 to 14.2] | 29.4 [10.3 to 56.0] | 16.7 [3.6 to 41.4] | 0 [0.0 to 16.8]
  Headache: Moderate | 12.0 [2.5 to 31.2] | 8.7 [1.1 to 28.0] | 4.2 [0.1 to 21.1] | 11.8 [1.5 to 36.4] | 16.7 [3.6 to 41.4] | 0 [0.0 to 16.8]
  Headache: Severe | 0 [0.0 to 13.7] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 19.5] | 0 [0.0 to 18.5] | 0 [0.0 to 16.8]
  Muscle pain: Mild | 16.0 [4.5 to 36.1] | 21.7 [7.5 to 43.7] | 0 [0.0 to 14.2] | 23.5 [6.8 to 49.9] | 33.3 [13.3 to 59.0] | 0 [0.0 to 16.8]
  Muscle pain: Moderate | 4.0 [0.1 to 20.4] | 17.4 [5.0 to 38.8] | 0 [0.0 to 14.2] | 0 [0.0 to 19.5] | 5.6 [0.1 to 27.3] | 0 [0.0 to 16.8]
  Muscle pain: Severe | 0 [0.0 to 13.7] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 19.5] | 0 [0.0 to 18.5] | 0 [0.0 to 16.8]
  Joint pain: Mild | 4.0 [0.1 to 20.4] | 4.3 [0.1 to 21.9] | 0 [0.0 to 14.2] | 0 [0.0 to 19.5] | 11.1 [1.4 to 34.7] | 0 [0.0 to 16.8]
  Joint pain: Moderate | 4.0 [0.1 to 20.4] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 19.5] | 0 [0.0 to 18.5] | 0 [0.0 to 16.8]
  Joint pain: Severe | 0 [0.0 to 13.7] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 19.5] | 0 [0.0 to 18.5] | 0 [0.0 to 16.8]
  Vomiting: Mild | 0 [0.0 to 13.7] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 5.9 [0.1 to 28.7] | 5.6 [0.1 to 27.3] | 10.0 [1.2 to 31.7]
  Vomiting: Moderate | 0 [0.0 to 13.7] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 19.5] | 0 [0.0 to 18.5] | 0 [0.0 to 16.8]
  Vomiting: Severe | 0 [0.0 to 13.7] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 19.5] | 0 [0.0 to 18.5] | 0 [0.0 to 16.8]
  Diarrhea: Mild | 4.0 [0.1 to 20.4] | 8.7 [1.1 to 28.0] | 4.2 [0.1 to 21.1] | 0 [0.0 to 19.5] | 5.6 [0.1 to 27.3] | 0 [0.0 to 16.8]
  Diarrhea: Moderate | 0 [0.0 to 13.7] | 0 [0.0 to 14.8] | 8.3 [1.0 to 27.0] | 0 [0.0 to 19.5] | 0 [0.0 to 18.5] | 0 [0.0 to 16.8]
  Diarrhea: Severe | 0 [0.0 to 13.7] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 19.5] | 0 [0.0 to 18.5] | 0 [0.0 to 16.8]

3. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Within 1 Month After Vaccination
Description: AE was defined as any untoward medical occurrence in clinical study participant, temporally associated with use of study intervention, whether or not considered related to study intervention. AEs included serious and all non-serious AE. SAEs were defined as AE that, at any dose: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability/incapacity; was congenital anomaly or birth defect; was suspected transmission via Pfizer product of infectious agent, pathogenic or nonpathogenic or was considered to be an important medical event. Only AEs collected by non-systematic assessment (i.e., excluding local reactions and systemic events) were included.
Time Frame: Within 1 month post Vaccination
Population: Safety population included all enrolled participants who received study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSVpreF 120 mcg: 5 to <18 Years [Healthy Participants] | RSVpreF 120 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 120 mcg: 2 to <5 Years | RSVpreF 60 mcg: 5 to <18 Years [Healthy Participants] | RSVpreF 60 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 60 mcg: 2 to <5 Years
Number analyzed (Participants) | 25 | 23 | 24 | 17 | 18 | 20
Percentage of participants | 0 [0.0 to 13.7] | 17.4 [5.0 to 38.8] | 12.5 [2.7 to 32.4] | 0 [0.0 to 19.5] | 27.8 [9.7 to 53.5] | 15.0 [3.2 to 37.9]

4. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) Throughout the Study
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. SAEs were defined as an AE that, at any dose: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability or incapacity; was a congenital anomaly or birth defect; was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or nonpathogenic or that was considered to be an important medical event.
Time Frame: Within 6 months post Vaccination
Population: Safety population included all enrolled participants who received study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSVpreF 120 mcg: 5 to <18 Years [Healthy Participants] | RSVpreF 120 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 120 mcg: 2 to <5 Years | RSVpreF 60 mcg: 5 to <18 Years [Healthy Participants] | RSVpreF 60 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 60 mcg: 2 to <5 Years
Number analyzed (Participants) | 25 | 23 | 24 | 17 | 18 | 20
Percentage of participants | 0 [0.0 to 13.7] | 4.3 [0.1 to 21.9] | 0 [0.0 to 14.2] | 0 [0.0 to 19.5] | 5.6 [0.1 to 27.3] | 0 [0.0 to 16.8]

5. Primary Outcome: Percentage of Participants Reporting Newly Diagnosed Chronic Medical Condition (NDCMCs) Throughout the Study
Description: An NDCMC was defined as a disease or medical condition, which was not previously identified, that was expected to be persistent or otherwise long-lasting in its effects.
Time Frame: Within 6 months post Vaccination
Population: Safety population included all enrolled participants who received study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSVpreF 120 mcg: 5 to <18 Years [Healthy Participants] | RSVpreF 120 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 120 mcg: 2 to <5 Years | RSVpreF 60 mcg: 5 to <18 Years [Healthy Participants] | RSVpreF 60 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 60 mcg: 2 to <5 Years
Number analyzed (Participants) | 25 | 23 | 24 | 17 | 18 | 20
Percentage of participants | 0 [0.0 to 13.7] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 19.5] | 0 [0.0 to 18.5] | 0 [0.0 to 16.8]

6. Secondary Outcome: Geometric Mean Titer of the Neutralizing Titers for RSV A and RSV B Before Vaccination and 1 Month After Vaccination
Description: Geometric mean titer (GMT) of neutralizing titers (NTs) of respiratory syncytial virus subgroup A and respiratory syncytial virus subgroup B (RSV A and RSV B) before vaccination and 1 month after vaccination were reported in this outcome measure. Assay results below the lower limit of quantification (LLOQ) were set to 0.5*LLOQ. GMTs and corresponding 2-sided CIs were calculated by exponentiating mean logarithm of titers and corresponding CIs (based on Student's t distribution).
Time Frame: Before vaccination and 1 month after vaccination
Population: Evaluable immunogenicity population (EIP) included all eligible participants who received the study intervention; had 1-month postvaccination blood collection 27 through 42 days after vaccination; had at least 1 valid and determinate assay result 1 month after vaccination; had no major protocol violations from vaccination through the 1-month postvaccination blood draw. Here, "Number Analyzed" signifies participants evaluable for the specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RSVpreF 120 mcg: 5 to <18 Years [Healthy Participants] | RSVpreF 120 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 120 mcg: 2 to <5 Years | RSVpreF 60 mcg: 5 to <18 Years [Healthy Participants] | RSVpreF 60 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 60 mcg: 2 to <5 Years
Number analyzed (Participants) | 24 | 21 | 24 | 15 | 18 | 20
Titer
  RSV A: Before vaccination: number analyzed (Participants) | 24 | 20 | 24 | 15 | 18 | 20
  RSV A: Before vaccination | 1168 [706 to 1932] | 2003 [1421 to 2823] | 529 [335 to 835] | 916 [653 to 1285] | 1667 [1035 to 2684] | 561 [309 to 1016]
  RSV A:1 Month after vaccination | 27862 [21493 to 36119] | 35503 [26876 to 46900] | 26146 [13301 to 51396] | 25341 [15394 to 41715] | 24053 [17440 to 33173] | 11004 [4287 to 28245]
  RSV B: Before vaccination: number analyzed (Participants) | 24 | 20 | 24 | 15 | 18 | 20
  RSV B: Before vaccination | 1206 [717 to 2027] | 1905 [1238 to 2930] | 391 [231 to 661] | 965 [668 to 1393] | 1760 [947 to 3272] | 499 [258 to 967]
  RSV B:1 Month after vaccination | 30251 [21607 to 42355] | 29019 [18786 to 44827] | 16504 [8267 to 32948] | 33351 [23565 to 47202] | 31174 [21756 to 44668] | 10659 [3526 to 32228]

7. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of the NTs for RSV A and RSV B From Before Vaccination to 1 Month After Vaccination
Description: GMFR of neutralizing titers of RSV A and RSV B from before vaccination to 1 month after vaccination were reported in this outcome measure. GMFR and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rises and the corresponding CIs (based on the Student's t distribution).
Time Frame: From before vaccination to 1 month after vaccination
Population: EIP included all eligible participants who received the study intervention; had 1-month postvaccination blood collection 27 through 42 days after vaccination; had at least 1 valid and determinate assay result 1 month after vaccination; had no major protocol violations from vaccination through the 1-month postvaccination blood draw. Here, ''Number of Participants Analyzed'' signifies participants evaluable of this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | RSVpreF 120 mcg: 5 to <18 Years [Healthy Participants] | RSVpreF 120 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 120 mcg: 2 to <5 Years | RSVpreF 60 mcg: 5 to <18 Years [Healthy Participants] | RSVpreF 60 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 60 mcg: 2 to <5 Years
Number analyzed (Participants) | 24 | 20 | 24 | 15 | 18 | 20
Fold rise
  RSV A | 21.9 [14.46 to 33.08] | 18.6 [13.03 to 26.55] | 42.8 [23.41 to 78.16] | 27.7 [17.81 to 42.93] | 13.9 [8.75 to 22.03] | 17.7 [9.02 to 34.67]
  RSV B | 24.4 [15.53 to 38.26] | 16.3 [9.91 to 26.83] | 39.8 [22.96 to 69.08] | 34.6 [21.63 to 55.23] | 17.0 [9.25 to 31.40] | 20.6 [10.00 to 42.50]

8. Secondary Outcome: Median Frequencies of RSV F Antigen-Specific Cluster of Differentiation 4 (CD4+) Thymus-Derived Lymphocytes (T) Cells Expressing Interferon (IFN) Gamma and Interleukin-4 (IL-4) Before Vaccination and 1 Month After Vaccination
Description: Median frequencies of RSV F antigen-specific CD4+ T cells expressing IFN gamma and IL-4 before vaccination and 1 month after vaccination were reported in this outcome measure. RSV F enzyme-linked immune absorbent spot assay (ELISpot) limit of detection (LOD) values were IFN gamma = 20 spot forming cell (SFC) per million peripheral blood mononuclear cell (PBMCs) and IL-4 = 4 SFC/million PBMCs. Assay results below LOD=0.5*LOD for analysis. Frequencies were defined as the count of the RSV F antigen-specific CD4+ T cells and median frequencies were defined as the median of the counts.
Time Frame: Before vaccination and 1 Month after vaccination
Population: EIP included all eligible participants who received the study intervention; had 1-month postvaccination blood collection 27 through 42 days after vaccination; had at least 1 valid and determinate assay result 1 month after vaccination; had no major protocol violations from vaccination through the 1-month postvaccination blood draw. Here, "Number of Participants Analyzed" = participants evaluable for this outcome measure and "Number Analyzed" = participants evaluable for specified rows.
Measure: Median (Full Range); unit: SFC/million PBMCs
Arm/Group | RSVpreF 120 mcg: 5 to <18 Years [Healthy Participants] | RSVpreF 120 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 120 mcg: 2 to <5 Years | RSVpreF 60 mcg: 5 to <18 Years [Healthy Participants] | RSVpreF 60 mcg: 5 to <18 Years [High Risk Participants] | RSVpreF 60 mcg: 2 to <5 Years
Number analyzed (Participants) | 23 | 21 | 22 | 15 | 18 | 17
SFC/million PBMCs
  INF gamma before vaccination: number analyzed (Participants) | 23 | 19 | 22 | 14 | 17 | 17
  INF gamma before vaccination | 47 [10 to 241] | 60 [10 to 193] | 10 [10 to 67] | 53 [10 to 277] | 41 [10 to 336] | 10 [10 to 79]
  INF gamma 1 month after vaccination: number analyzed (Participants) | 22 | 21 | 21 | 15 | 18 | 17
  INF gamma 1 month after vaccination | 255 [10 to 829] | 293 [10 to 1339] | 61 [10 to 257] | 244 [23 to 1027] | 187 [10 to 780] | 45 [10 to 184]
  IL-4 before vaccination: number analyzed (Participants) | 23 | 19 | 22 | 14 | 17 | 17
  IL-4 before vaccination | 2 [2 to 2] | 2 [2 to 11] | 2 [2 to 2] | 2 [2 to 4] | 2 [2 to 5] | 2 [2 to 4]
  IL-4 1 month after vaccination: number analyzed (Participants) | 22 | 21 | 21 | 15 | 18 | 17
  IL-4 1 month after vaccination | 2 [2 to 16] | 4 [2 to 28] | 2 [2 to 7] | 2 [2 to 24] | 2 [2 to 15] | 2 [2 to 13]

ADVERSE EVENTS:
Time Frame: Local reactions and systemic events: Within 7 days after vaccination. SAEs: Within 6 months post Vaccination and other AEs: Within 1 month post Vaccination
Description: Same event may appear as both non-SAE and SAE but what is presented are distinct events. An event may be categorized as serious in one participant and nonserious in another participant or one participant may have experienced both serious and non-serious event. Safety population included all enrolled participants who received study intervention.
Groups:
- Healthy RSVpreF 120 Micrograms (mcg): Healthy participants with 5 to < 18 years of age received a single dose of 120 mcg RSVpreF as standard dose level intramuscularly into the deltoid muscle (Vaccination 1) on Day 1.
- High Risk RSVpreF 120 mcg: High risk participants with 5 to < 18 years of age received a single dose of 120 mcg RSVpreF as standard dose level intramuscularly into the deltoid muscle (Vaccination 1) on Day 1.
- 2 to < 5 Years RSVpreF 120 mcg: Participants with 2 to < 5 years of age received a single dose of 120 mcg RSVpreF as standard dose level intramuscularly into the deltoid muscle (Vaccination 1) on Day 1.
- Healthy RSVpreF 60 mcg: Healthy participants with 5 to < 18 years of age received a single dose of 60 mcg RSVpreF as standard dose level intramuscularly into the deltoid muscle (Vaccination 1) on Day 1.
- High Risk RSVpreF 60 mcg: High risk participants with 5 to < 18 years of age received a single dose of 60 mcg RSVpreF as standard dose level intramuscularly into the deltoid muscle (Vaccination 1) on Day 1.
- 2 to < 5 Years RSVpreF 60 mcg: Participants with 2 to < 5 years of age received a single dose of 60 mcg RSVpreF as standard dose level intramuscularly into the deltoid muscle (Vaccination 1) on Day 1.
Arm/Group | Healthy RSVpreF 120 Micrograms (mcg) | High Risk RSVpreF 120 mcg | 2 to < 5 Years RSVpreF 120 mcg | Healthy RSVpreF 60 mcg | High Risk RSVpreF 60 mcg | 2 to < 5 Years RSVpreF 60 mcg
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23 | 0/24 | 0/17 | 0/18 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/23 | 0/24 | 0/17 | 1/18 | 0/20
Other Adverse Events (participants affected / at risk) | 17/25 | 15/23 | 9/24 | 12/17 | 14/18 | 13/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy RSVpreF 120 Micrograms (mcg) (N=25) | High Risk RSVpreF 120 mcg (N=23) | 2 to < 5 Years RSVpreF 120 mcg (N=24) | Healthy RSVpreF 60 mcg (N=17) | High Risk RSVpreF 60 mcg (N=18) | 2 to < 5 Years RSVpreF 60 mcg (N=20)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy RSVpreF 120 Micrograms (mcg) (N=25) | High Risk RSVpreF 120 mcg (N=23) | 2 to < 5 Years RSVpreF 120 mcg (N=24) | Healthy RSVpreF 60 mcg (N=17) | High Risk RSVpreF 60 mcg (N=18) | 2 to < 5 Years RSVpreF 60 mcg (N=20)
Headache (HEADACHE) (Nervous system disorders) | 7 (7) | 8 (8) | 1 (1) | 7 (7) | 6 (6) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Vomiting (VOMITING) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Erythema (REDNESS) (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 5 (5) | 9 (9) | 0 (0) | 4 (4) | 7 (7) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (FATIGUE) (General disorders) | 8 (8) | 10 (10) | 7 (7) | 8 (8) | 9 (9) | 7 (7)
Injection site erythema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site pain (PAIN AT INJECTION SITE) (General disorders) | 12 (12) | 11 (11) | 2 (2) | 7 (7) | 10 (10) | 3 (3)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (FEVER) (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Swelling (SWELLING) (General disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2024-02-11): https://cdn.clinicaltrials.gov/large-docs/54/NCT05900154/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/54/NCT05900154/SAP_001.pdf